CLINICAL TRIAL: NCT05957458
Title: Retrospective Study of Photobiomodulation Therapy on Myopia Control With Airdoc Red Light at Wavelength of 650nm
Brief Title: Myopia Control With Three Lever Irradiance of PBM Therapy in Children and Adults
Acronym: MCPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Airdoc Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Airdoc MPC Co.Ltd.
Record Dates: First submitted 2023-05-23; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Myopia; Amblyopia; Refractive Error - Myopia Axial; Ametropia
Keywords: Myopia; PBM therapy; LLLT
MeSH Terms: conditions — Myopia; Amblyopia; Refractive Errors | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Three groups are all treated with PBM therapy with follow-up but they irradiance is different while one group is as the control.
Masking Description: No mask for all. Open and retrospective study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moderate irradiance of PBM therapy to myopia (Experimental): The PBM therapy irradiance is about 0.60mW. It is asked subjects to look at the light binocularly with fusion through the pupils with natural pupils. The distance between the light and the pupils is about 5~10cm. The treatment of each session is 3 minutes and twice daily administration while the interval time between two session is equal or larger than 4 hours with twice daily administration.
  Interventions: Device: Airdoc device of red light for Myopia
- Extra low irradiance PBM therapy group (Sham Comparator): The PBM therapy irradiance is about 0.37mW. It is asked subjects to look at the light binocularly with fusion through the pupils with natural pupils. The distance between the light and the pupils is about 5~10cm. The treatment of each session is 3 minutes and twice daily administration while the interval time between two session is equal or larger than 4 hours with twice daily administration.
  Interventions: Device: Airdoc device of red light for Myopia
- high lever PBM therapy group (Experimental): The PBM therapy irradiance is about 1.20mW. It is asked subjects to look at the light binocularly with fusion through the pupils with natural pupils. The distance between the light and the pupils is about 5~10cm. The treatment of each session is 3 minutes and twice daily administration while the interval time between two session is equal or larger than 4 hours with twice daily administration.
  Interventions: Device: Airdoc device of red light for Myopia
- Control (No Intervention): Without PBM therapy group.

INTERVENTIONS:
Device: Airdoc device of red light for Myopia — This light is Narrow-Band, Long-Wavelength Lighting with three different illumination (400lux, 800lux, 1200lux) or irridiance (1.2mW, 0.6mW, 0.37mW) respectively. And the wavelength is 650nm. It allows biocular therapy.
  Other Names: low lever laser therapy; photobiomodulation therapy; low lever light therapy
  Arms: Extra low irradiance PBM therapy group; Moderate irradiance of PBM therapy to myopia; high lever PBM therapy group

SUMMARY:
Photobiomodulation therapy, that is, Low-level red-light technology provides a new and innovative myopia control approach. This strategy enables relatively high energies of light to be delivered at much shorter durations of exposure to induce the myopia control effect. The efficacy of the low-level red-light technology has been proven in a Chinese populationb for the recent 3 years with evidence based papers and amazing results. However, there's not yet evidence to demonstrate the relationship between the dose response effect of photobiomodulation therapy on myopia control at the different age lever.

DETAILED DESCRIPTION:
Previous trial has demonstrated that 3-minutes per session twice a day repeated low-level red-light treatment at the irridiance of 2.3mW（2.0~2.5mW) controlled 87.7% of refraction progression and 76.8% of axial length elongation when the time of compliance to the treatment was 75%. Retrospective analyze other irriadance of 1.2mW, 0.6mW and 0.37mW culturally diverse groups will confirm and translate this technology into a solution for myopia control globally.

ELIGIBILITY:
Inclusion Criteria:

* Myopia or near Myopia with younger age
* Without other intervention of myopia control, including atropine, Misight contact lens, special design lens to control myopia, orthokeratology and other red light devices.
* Follow-up at least once
* With baseline data of ocular parameters before the follow-up

Exclusion Criteria:

* Photophobia
* Allergy to red light
* Severe ocular progressing diseases or systemic diseases
* The data is unacceptable with reasonable explanations

Ages: 4 Years to 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Axial length shortening comparing to that value of baseline (mm） | 12-month
  Measured with optial coherent methods with the same device assistant with the same techinician
Axial length shortening comparing to that value of baseline (mm） | 1-month
  Measured with optial coherent methods with the same device assistant with the techinician
Axial length shortening comparing to that value of baseline (mm） | 6-month
  Measured with optial coherent methods with the same device assistant with the same techinician

SECONDARY OUTCOMES:
Refractive changes at the follow-up from the baseline (D) | 12-month
  Spherical Equivalence were recorded with the right eyes only

CONTACTS AND LOCATIONS:
Overall Officials: QIU JENNY, MD, Principal Investigator — Airdoc MPC Co, Ltd.
Locations (1):
- Qiu Jenny, Beijing, Haidian District, China

REFERENCES:
- [Background] Zhou L, Tong L, Li Y, Williams BT, Qiu K. Photobiomodulation therapy retarded axial length growth in children with myopia: evidence from a 12-month randomized controlled trial evidence. Sci Rep. 2023 Feb 27;13(1):3321. doi: 10.1038/s41598-023-30500-7. PMID 36849626